CLINICAL TRIAL: NCT00418457
Title: Regional Anesthesia and Breast Cancer Recurrence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, d sessler, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 06-692
Record Dates: First submitted 2007-01-03; First posted 2007-01-04 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Breast Neoplasms
Keywords: Breast Cancer; Anesthesia; regional; cancer recurrence; Anesthesia; inhalational; Analgesia; opioid
MeSH Terms: conditions — Breast Neoplasms; Agnosia | interventions — Anesthesia, General; Analgesics, Opioid; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- General anesthesia and opioid (Active Comparator): General anesthesia followed by opioid administration
  Interventions: Drug: General anesthesia and opioids
- Regional analgesia and propofol (Active Comparator): Regional anesthesia and analgesia (either epidural or paravertebral) combined with propofol
  Interventions: Drug: Regional analgesia and propofol

INTERVENTIONS:
Drug: General anesthesia and opioids — General anesthesia, usually with sevoflurane, and opioid analgesia
  Other Names: General anesthesia
  Arms: General anesthesia and opioid
Drug: Regional analgesia and propofol — Regional anesthesia and analgesia (either epidural or paravertebral), combined with deep sedation or general anesthesia
  Other Names: Regional analgesia
  Arms: Regional analgesia and propofol

SUMMARY:
In this multi-center trial, Stage 1-3 patients having mastectomies or isolated lumpectomy with axillary node dissection will be randomly assigned to thoracic epidural or paravertebral anesthesia/analgesia, or to general anesthesia and morphine analgesia. Participants will be followed for up to 10 years to determine the rate of cancer recurrence or metastasis.

DETAILED DESCRIPTION:
Surgery is the primary and most effective treatment of breast cancer, but residual disease in the form of scattered micrometastases and tumor cells are usually unavoidable. Whether minimal residual disease results in clinical metastases is a function of host defense and tumor survival and growth. At least three perioperative factors shift the balance toward progression of minimal residual disease:

1. Surgery per se depresses cell-mediated immunity, reduces concentrations of tumor-related anti-angiogenic factors (e.g., angiostatin and endostatin), increases concentrations of pro-angiogenic factors such as VEGF, and releases growth factors that promote local and distant growth of malignant tissue.
2. Anesthesia impairs numerous immune functions, including those of neutrophils, macrophages, dendritic cells, T-cell, and natural killer cells.
3. Opioid analgesics inhibit both cellular and humoral immune function in humans, increase angiogenesis, and promote breast tumor growth in rodents.

However, regional analgesia attenuates or prevents each of these adverse effects by largely preventing the neuroendocrine surgical stress response, eliminating or reducing the need for general anesthesia, and minimizing opioid requirement. Animal studies indicate that regional anesthesia and optimum postoperative analgesia independently reduce the metastatic burden in animals inoculated with breast adenocarcinoma cells following surgery. Preliminary data in cancer patients are also consistent: paravertebral analgesia for breast cancer surgery reduced risk of recurrence or metastasis approximately four-fold (95% CI of estimated hazard ratio is 0.71 - 0.06) during a 2.5 to 4-year follow-up period compared to opioid analgesia. The investigators will thus test the hypothesis that recurrence after breast cancer surgery is lower with regional anesthesia/analgesia than with general anesthesia and opioid analgesia.

In this multi-center trial, Stage 1-3 patients having mastectomies will be randomly assigned to thoracic epidural or paravertebral anesthesia/analgesia, or to general anesthesia and opioid analgesia. As with all time-to-event trials, interim and final analyses are based on the number of outcome events (recurrences in this case) rather than enrollment. The number of patients required is just an estimate and varies based on actual recurrence rates which in turn depend on patients' stage and grade, and ancillary treatments. There will be three evenly spaced interim analyses and a final analysis at 351 recurrences. Confirming our hypothesis will indicate that a minor modification to anesthetic management, one that can be implemented with little risk or cost, will reduce the risk of cancer recurrence - a complication that is often ultimately lethal.

ELIGIBILITY:
Inclusion Criteria:

* Primary breast cancer without known extension beyond the breast and axillary nodes (i.e. believed to be Tumor Stage 1-3, Nodes 0-2)
* Scheduled for unilateral or bilateral mastectomy with or without implant (isolated "lumpectomy" will not qualify)
* Isolated "lumpectomy" with axillary node dissection (anticipated removal of at least five nodes)
* Written informed consent, including willingness to be randomized to morphine or regional analgesia

Exclusion Criteria:

* Previous surgery for breast cancer (except diagnostic biopsies)
* Inflammatory breast cancer
* Age < 18 or > 85 years old
* Scheduled free flap reconstruction
* ASA Physical Status ≥ 4
* Any contraindication to epidural or paravertebral anesthesia and analgesia (including coagulopathy, abnormal anatomy)
* Any contraindication to midazolam, propofol, sevoflurane, fentanyl, or morphine
* Other cancer not believed by the attending surgeon to be in long-term remission
* Systemic disease believed by the attending surgeon to present ≥ 25% two-year mortality

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2108 (Actual)
Dates: Start 2007-01; Primary Completion 2018-02 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Sessler, MD, Principal Investigator — The Cleveland Clinic
Locations (6):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States
- Medical University of Vienna, Vienna, Austria
- Peking Union Medical College Hospital, Beijing, China
- University of Düsseldorf, Düsseldorf, Germany
- Mater Misericordiae Hospital, Dublin, Ireland
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li M, Zhang Y, Pei L, Zhang Z, Tan G, Huang Y. Potential Influence of Anesthetic Interventions on Breast Cancer Early Recurrence According to Estrogen Receptor Expression: A Sub-Study of a Randomized Trial. Front Oncol. 2022 Feb 10;12:837959. doi: 10.3389/fonc.2022.837959. eCollection 2022. PMID 35223519
- [Derived] Aghamelu O, Buggy P, Smith G, Inzitari R, Wall T, Buggy DJ. Serum NETosis expression and recurrence risk after regional or volatile anaesthesia during breast cancer surgery: A pilot, prospective, randomised single-blind clinical trial. Acta Anaesthesiol Scand. 2021 Mar;65(3):313-319. doi: 10.1111/aas.13745. Epub 2020 Nov 29. PMID 33187020
- [Derived] Sessler DI, Pei L, Huang Y, Fleischmann E, Marhofer P, Kurz A, Mayers DB, Meyer-Treschan TA, Grady M, Tan EY, Ayad S, Mascha EJ, Buggy DJ; Breast Cancer Recurrence Collaboration. Recurrence of breast cancer after regional or general anaesthesia: a randomised controlled trial. Lancet. 2019 Nov 16;394(10211):1807-1815. doi: 10.1016/S0140-6736(19)32313-X. Epub 2019 Oct 20. PMID 31645288
- [Derived] Levins KJ, Prendeville S, Conlon S, Buggy DJ. The effect of anesthetic technique on micro-opioid receptor expression and immune cell infiltration in breast cancer. J Anesth. 2018 Dec;32(6):792-796. doi: 10.1007/s00540-018-2554-0. Epub 2018 Sep 18. PMID 30229370
- [Derived] Kim R. Anesthetic technique and cancer recurrence in oncologic surgery: unraveling the puzzle. Cancer Metastasis Rev. 2017 Mar;36(1):159-177. doi: 10.1007/s10555-016-9647-8. PMID 27866303
- [Derived] Pei L, Zhou Y, Tan G, Mao F, Yang D, Guan J, Lin Y, Wang X, Zhang Y, Zhang X, Shen S, Xu Z, Sun Q, Huang Y; Outcomes Research Consortium. Ultrasound-Assisted Thoracic Paravertebral Block Reduces Intraoperative Opioid Requirement and Improves Analgesia after Breast Cancer Surgery: A Randomized, Controlled, Single-Center Trial. PLoS One. 2015 Nov 20;10(11):e0142249. doi: 10.1371/journal.pone.0142249. eCollection 2015. PMID 26588217
- [Derived] Wu J, Buggy D, Fleischmann E, Parra-Sanchez I, Treschan T, Kurz A, Mascha EJ, Sessler DI. Thoracic paravertebral regional anesthesia improves analgesia after breast cancer surgery: a randomized controlled multicentre clinical trial. Can J Anaesth. 2015 Mar;62(3):241-51. doi: 10.1007/s12630-014-0285-8. Epub 2014 Dec 6. PMID 25480319
- [Derived] Jaura AI, Flood G, Gallagher HC, Buggy DJ. Differential effects of serum from patients administered distinct anaesthetic techniques on apoptosis in breast cancer cells in vitro: a pilot study. Br J Anaesth. 2014 Jul;113 Suppl 1:i63-7. doi: 10.1093/bja/aet581. Epub 2014 Jul 9. PMID 25009197
- [Derived] Buckley A, McQuaid S, Johnson P, Buggy DJ. Effect of anaesthetic technique on the natural killer cell anti-tumour activity of serum from women undergoing breast cancer surgery: a pilot study. Br J Anaesth. 2014 Jul;113 Suppl 1:i56-62. doi: 10.1093/bja/aeu200. Epub 2014 Jul 9. PMID 25009196

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | General Anesthesia and Opioid | Regional Analgesia and Propofol
Started | 1065 | 1043
Completed | 1065 | 1043
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | General Anesthesia and Opioid | Regional Analgesia and Propofol | Total
Number analyzed (Participants) | 1065 | 1043 | 2108
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (11) | 53 (12) | 53 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1065 | 1043 | 2108
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 989 | 972 | 1961
  Unknown or Not Reported | 72 | 68 | 140

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Breast Cancer Recurrence After Breast Cancer Surgery
Description: time to breast cancer recurrence from the end of surgery.
Time Frame: up to 10 years
Measure: Number; unit: participants
Arm/Group | General Anesthesia and Opioid | Regional Analgesia and Propofol
Number analyzed (Participants) | 1065 | 1043
participants | 111 | 102
Statistical Analysis 1: Comparison: General Anesthesia and Opioid vs Regional Analgesia and Propofol; Test type: Superiority; p = 0.84, Regression, Cox; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.74 to 1.28]

2. Secondary Outcome: Number of Participants That Experienced Post-Surgical Pain
Description: Brief Pain Inventory is used to evaluate with values of any pain vs. no pain (binary)
Time Frame: 6 months and 1 year
Population: data was not available/collected for all participants due to lost follow up or miss phone call.
Measure: Count of Participants; unit: Participants
Arm/Group | General Anesthesia and Opioid | Regional Analgesia and Propofol
Number analyzed (Participants) | 872 | 856
Participants
  at 6-month | 456 | 442
  1-year: number analyzed (Participants) | 852 | 854
  1-year | 232 | 239
Statistical Analysis 1: Comparison: General Anesthesia and Opioid vs Regional Analgesia and Propofol; Test type: Superiority; p = 0.70, GEE; Odds Ratio (OR) = 1, 95% CI 2-sided [0.85 to 1.17]

3. Secondary Outcome: Number of Participants That Experienced Neuropathic Pain After Surgery
Description: neuropathic pain is a binary outcome: any pain vs. no pain
Time Frame: 6 month and 1 year
Population: data was not available/collected for all participants due to lost follow up or miss phone call.
Measure: Count of Participants; unit: Participants
Arm/Group | General Anesthesia and Opioid | Regional Analgesia and Propofol
Number analyzed (Participants) | 870 | 859
Participants
  at 6-month | 89 | 87
  1-year: number analyzed (Participants) | 854 | 857
  1-year | 57 | 57
Statistical Analysis 1: Comparison: General Anesthesia and Opioid vs Regional Analgesia and Propofol; Test type: Superiority; p = 0.81, GEE; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.75 to 1.28]

4. Secondary Outcome: SF-12 PCS Score
Description: Physical and Mental Health Composite Scores (PCS & MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: 6 month and 1 year
Population: data was not available/collected for all participants due to lost follow up or miss phone call.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | General Anesthesia and Opioid | Regional Analgesia and Propofol
Number analyzed (Participants) | 804 | 807
score on a scale
  at 6-month: number analyzed (Participants) | 804 | 788
  at 6-month | 49.7 (8.1) | 49.8 (8.2)
  1-year: number analyzed (Participants) | 800 | 807
  1-year | 52.3 (6.7) | 52.1 (7.3)
Statistical Analysis 1: Comparison: General Anesthesia and Opioid vs Regional Analgesia and Propofol; Test type: Superiority; p = 0.96, Mixed Models Analysis; Mean Difference (Final Values) = -0.014, 95% CI 2-sided [-0.63 to 0.60]

5. Secondary Outcome: SF-12 MCS Score
Description: as for outcome 4
Time Frame: 6 month and 1 year
Population: data was not available/collected for all participants due to lost follow up or miss phone call.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | General Anesthesia and Opioid | Regional Analgesia and Propofol
Number analyzed (Participants) | 804 | 807
units on a scale
  at 6-month: number analyzed (Participants) | 800 | 807
  at 6-month | 48.1 (8.6) | 48.7 (8.1)
  1-year: number analyzed (Participants) | 804 | 788
  1-year | 48 (9.7) | 48.7 (9.4)
Statistical Analysis 1: Comparison: General Anesthesia and Opioid vs Regional Analgesia and Propofol; Test type: Superiority; p = 0.043, Mixed Models Analysis; Mean Difference (Final Values) = 0.75, 95% CI 2-sided [0.02 to 1.48]

ADVERSE EVENTS:
Time Frame: UP to 10 years After surgery
Arm/Group | General Anesthesia and Opioid | Regional Analgesia and Propofol
All-Cause Mortality (participants affected / at risk) | 22/1065 | 18/1043
Serious Adverse Events (participants affected / at risk) | 0/1065 | 0/1043
Other Adverse Events (participants affected / at risk) | 0/1065 | 0/1043

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/57/NCT00418457/Prot_SAP_000.pdf